CLINICAL TRIAL: NCT02078141
Title: Monocentric, Prospective, Uncontrolled Pilot Study of Extra Cardiomyocytary Fixation Profile in 18F-fluorodeoxyglucose (FDG) Positron Emission Tomography in Patients With Dilated Cardiomyopathy.
Brief Title: 18F-deoxyglucose (FDG) PET-CMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC14_0002
Record Dates: First submitted 2014-02-21; First posted 2014-03-05 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Patients With Idiopathic Dilated Cardiomyopathy
Keywords: 18F-deoxyglucose (FDG) PET, idiopathic Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-deoxyglucose (FDG) (Experimental): 18F-deoxyglucose (FDG)
  Interventions: Drug: 18F-deoxyglucose (FDG)

INTERVENTIONS:
Drug: 18F-deoxyglucose (FDG) — 18F-deoxyglucose (FDG) One injection of 3.5 MBq/kg of 18FDG with a minimum of 220 MBq and a maximum of 400 MBq

SUMMARY:
18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) may have application in a promising tool for identification of myocardial inflammation in patients with dilated cardiomyopathy (DCM).Therefore, the purpose of the study is to confirm the hypothesis of the fixation of FDG in non cardiomyocyte cells in a number of patients with DCM, to specify the frequency and describe the different binding profiles in comparison with MRI data.

Patients will perform an ethologic evaluation of a non ischemic DCM with in a cardiac MRI.

All patients will have with in 4 weeks after the MRI a 18F-fluorodeoxyglucose (FDG) PET. A high fat and low carbohydrate diet and an heparin injection will be prescribed to patients before this FDG PET.

Patients will be identified as FDG+ or FDG -. The clinical status of the patient will be completed by a 12 months evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age
* Patients with DCM as defined by the European Society of Cardiology and recognized as such by the clinician cardiologist
* DCM diagnosed for more than two weeks without new ventricular arrhythmias or AuriculoVentricular Block (AVB) second or third degree , who responded to the usual treatment in the first two weeks of treatment
* No family history of DCM
* Lake of clinical or biological cases for periphiral myopathy or myotonia
* Absence of other causes of non-family DCM discovered during the initial etiological ( some deficiency , toxic alcoholic or drug )
* Patients who underwent cardiac MRI for etiological DCM for less than four weeks at the time of obtaining consent
* Patients who have read and understood the information letter and who signed the consent form
* Affiliated to a social insurance

Exclusion Criteria:

* Ischemic cardiomyopathy defined by history of myocardial infarction or myocardial revascularization , stenosis ≥ 75% of the core or the left coronary artery anterior interventricular proximal stenosis ≥ 75% on at least two epicardial vessels
* Significant organic valvular echocardiography
* Eosinophilia or immuno- allergic mechanism suspected
* History of acute myocarditis
* History of sarcoidosis
* Family history of DCM
* History of chemotherapy with anthracyclines
* Patient with signs of circulatory failure or congestive heart failure requiring intravenous positive inotropic therapy or diuretic therapy
* Treatment immunosuppressive received from cardiac MRI
* Hypersensitivity to heparin.
* History of severe thrombocytopenia type II ( heparin induced thrombocytopenia or immuno- allergic thrombocytopenia ) , heparin or unfractionated heparin , low molecular weight
* Other causes of non-family DCM discovered during the initial etiological ( some deficiency , toxic alcohol or medication , endocrine )
* Patients with active neoplasia
* Patients with chronic liver disease
* Patients with connective : rheumatoid arthritis , systemic lupus erythematosus , systemic sclerosis , dermato- polymyositis , mixed connective
* Patients with Crohn's disease
* Patients with active tuberculosis
* Pregnant or lactating women
* Minors
* Major Trust
* No affiliation to a social insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Determine the percentage of patients with a diagnostic potential of the 18F-FDG PET in the detection of a significant non-cardiomyocyte hypermetabolism | 12 months
  We want to objective a significant hypermetabolic extra-cardiomyocyte by 18F-FDG PET examination, in favor of myocardial inflammation in patients with DCM diagnosed for more than two weeks without new ventricular arrhythmias or second AVB or third degree, and who responded to the usual treatment in the first two weeks of treatment.

SECONDARY OUTCOMES:
Comparison of clinical, biology, and left and ventricular remodeling at the time of diagnosis of DCM between the group of patients with significative myocardial no cardiomyocytaire uptake (FDG +) and those with no uptake (FDG -) | 12 months
Evaluate the performance of 18F-FDG PET for the detection of myocardial inflammation in the initial evaluation of DCM patients compared to cardiac MRI | 12 months
Describe the different profile of FDG fixation within the group of patients FDG + | 12 months
impact of the presence or absence of a non-cardiomyocyte uptake of 18F-FDG PET at diagnosis of DCM in regard to the clinical status, ultrasound and MRI results | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Piriou, MD, Principal Investigator — Nantes UH
Locations (2):
- France (2):
  - Nantes UH, Nantes
  - West Cancerology Institute/Nantes UH : PET plateform, Saint-Herblain